CLINICAL TRIAL: NCT04392739
Title: A Post Marketing Study of the Safety, Tolerability, and Pharmacokinetics of TPOXX In Adult Subjects Weighing More Than 120 KG
Brief Title: Safety, Tolerability and PK of TPOXX in Adults Weighing More Than 120 KG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SIGA-246-022
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — tecovirimat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPOXX (Other): TPOXX 600 mg BID x 7 days
  Interventions: Drug: Tpoxx

INTERVENTIONS:
Drug: Tpoxx — oral antiviral

SUMMARY:
Safety and PK study in adults weighing more than 120 kg

DETAILED DESCRIPTION:
The primary objective of this study is to determine the pharmacokinetic (PK) profile of 600 mg oral TPOXX (3 × 200-mg capsules) administered twice daily (BID) for 7 days in adult subjects weighing more than 120 kg to determine if a change in dosing regimen would be needed in these patients.

Secondary:

The secondary objective of this study is to evaluate the safety and tolerability of 600 mg oral TPOXX administered BID for 7 days in healthy adult subjects weighing more than 120 kg.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18 and 50 years of age, inclusive.
2. Subject has a body weight >120 kg at screening, at check-in on Day -1, and prior to dosing on Day 1.
3. Women of childbearing potential, have a negative β human chorionic gonadotropin pregnancy test (serum) at the screening visit and a confirmatory negative serum pregnancy test on Day -1 before receipt of study drug, and meet 1 of the following criteria:

   1. The subject or their partner has undergone surgical sterilization
   2. The subject is postmenopausal, defined as 12 consecutive months with no menses without an alternative medical cause and has a documented plasma follicle-stimulating hormone level >40 IU/mL
   3. The subject agrees to be abstinent (ie, heterosexually inactive or women in a religious order)
   4. The subject agrees to consistently use 1 of the following methods of contraception from the beginning of screening (which they had been consistently using for at least 30 days before the first dose of study drug) through 30 days after the last dose of study drug:

   i. Condoms, male or female, with a spermicide NOTE: For male subjects, condoms must be used for 90 days after the last dose of study drug.

   ii. Diaphragm or cervical cap with spermicide

   iii. Intrauterine device with spermicide

   iv. Oral contraceptives or other hormonal methods NOTE: Subject must agree to use an additional nonhormonal method of contraception in conjunction with oral contraceptives.

   v. Male sexual partner who had undergone a vasectomy at least 3 months before screening
4. Male subjects must agree to not donate sperm from the first dose of study drug through 90 days after the last dose of study drug.
5. Subject is considered by the investigator to be in good general health as determined by medical history (no hospitalizations for chronic medical conditions in the previous 2 years), clinical laboratory results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at screening.
6. Subject agrees to comply with all protocol requirements.
7. Subject is able to provide written informed consent.
8. Subject agrees to comply with the dietary requirements.
9. Subject does not intend to lose

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subject is a female who is pregnant or breastfeeding or planning to become pregnant within 3 months after the last dose of study drug.
2. Subject has a history of any clinically significant conditions including:

   * Asthma treated with oral systemic steroids within the past 6 months
   * Diabetes mellitus (type 1 or 2), with the exception of gestational diabetes
   * Thyroidectomy or thyroid disease that required medication within the past 12 months
   * Serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years
   * Head trauma resulting in a diagnosis of traumatic brain injury other than concussion
   * Frequent episodes of headache.
3. Subject has received treatment in another clinical study of an investigational drug (or medical device) within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug.
4. Subject has been previously enrolled in any clinical study involving TPOXX (tecovirimat).
5. Subject has a history of relevant drug and/or food allergies (ie, allergy to tecovirimat or excipients, or any significant food allergy that could preclude a standard diet in the study site).
6. Subject has any condition possibly affecting drug absorption (eg, previous surgery on the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gallbladder, or pancreas, with the exception of appendectomy).
7. Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of the first dose of study drug), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to these criteria (eg, stable, mild joint disease unassociated with collagen vascular disease) may be made following discussions with the medical monitor.

   Page 10
8. Subject has a history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or risk factors for torsades de pointes (eg, heart failure, hypokalemia).
9. Subject has a family history of sudden cardiac death, not clearly due to acute myocardial infarction.
10. Subject has a seizure disorder or history of seizures (does not include childhood febrile seizures) or a past history that increases seizure risks such as significant head injury that caused loss of consciousness or other changes in the subject's daily function, concussion, stroke, central nervous system infection or disease, or alcohol or drug abuse or family history of idiopathic seizures.
11. Subject has a history of a peptic ulcer or significant gastrointestinal bleed.
12. Subject has a bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with blood draws.
13. Subject has a malignancy that is active, or treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that is likely to recur during the period of the study (subject should be in complete remission for at least 5 years).
14. Subject has neutropenia or other blood dyscrasia determined to be clinically significant by the investigator.
15. Subject has used any of the following prohibited medications from within 7 days (or 5 half-lives, whichever is longer) before the first dose of study drug: antidiabetic medication; anticoagulants; anticonvulsants; substrates of the breast cancer resistance protein transporter including methotrexate, mitoxantrone, imatinib, irinotecan, lapatinib, rosuvastatin, sulfasalazine, and topotecan; substrates of CYP2C8 including repaglinide, paclitaxel, Montelukast, pioglitazone, rosiglitazone; and substrates of CYP2C19 including S-mephenytoin, clobazam, diazepam, rabeprazole, voriconazole, lansoprazole, and omeprazole. Medications not listed here that are known (or thought) to be CYP3A4 substrates may be allowed at the investigator's discretion, after consultation with the medical monitor, if administration poses little to no risk to the subject.
16. Subject has a history of drug or alcohol abuse or dependency within the last year before screening.
17. Subject has a history of an eating disorder.
18. Subject has a current or recent (<30 days before screening) history of clinically significant bacterial, fungal, or mycobacterial infection.
19. Subject has a current clinically significant viral infection.
20. Subject has a known clinically significant chronic viral infection (eg, human T cell lymphotropic virus I or II).
21. Subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or caffeine- or xanthine-containing products within 48 hours before the first dose of study drug or throughout the study.
22. Subject has used any prescription (excluding hormonal birth control) or over-the-counter medication (including herbal or nutritional supplements) within 14 days before the first dose of study drug.
23. Subject demonstrates long-term use (≥14 consecutive days) of glucocorticoids including oral or parenteral prednisone or equivalent (>20 mg total dose per day) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 1 month (low-dose [≤800 mcg/day of beclomethasone dipropionate or equivalent] inhaled and topical steroids are allowed).
24. Subject has donated >450 mL blood or blood components within 30 days before the first dose of study drug. The investigator should instruct subjects who participate in this study to not donate blood or blood components for 4 weeks after the completion of the study.
25. Subject is a smoker or has used nicotine or nicotine-containing products (eg, cigarettes, electronic vapor cigarettes, cigars, chewing tobacco, snuff, nicotine patches, or nicotine gum) within 6 months before the first dose of study drug.
26. Subject has consumed pomegranate or pomegranate juice, pomelo fruits or pomelo juice, or alcohol within 72 hours before the first dose of study drug.
27. Subject reports participation in strenuous activity or contact sports within 24 hours before the first dose of study drug.
28. Subject has known hepatitis B or C infection or positive test for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus type 1 or 2 antibodies at screening.
29. Subject has a positive test result for amphetamines (including methamphetamines and ecstasy/methylenedioxymethamphetamine), barbiturates, benzodiazepines, cannabinoids (including tetrahydrocannabinol), cocaine metabolites, opiates (including heroin, codeine, and oxycodone), or alcohol at screening or check-in.
30. Subject has any of the following laboratory test results within 28 days before the first dose of study drug:

    * Estimated serum creatinine clearance (Cockcroft-Gault) <90 mL/min
    * Creatinine in males >1.7 mg/dL and in females >1.4 mg/dL (1.3 times the upper central laboratory reference range)
    * Hemoglobin ≤10% of the lower central laboratory reference range
    * White blood cell count not within the central laboratory reference range
    * Absolute neutrophil count <1000 cells/mm3
    * Platelets not within ±10% of central laboratory reference range
    * Alanine aminotransferase >1.5 times above the upper central laboratory reference range
    * Aspartate aminotransferase >1.5 times above the upper central laboratory reference range
    * Alkaline phosphatase >20% above the upper central laboratory reference range
    * Hemoglobin A1c ≥7.0%
    * Cholesterol ≥300 mg/dL and low-density lipoprotein ≥190 mg/dL.
31. Subject has a blood pressure considered to be clinically significant by the investigator. Blood pressure may be retested twice in the sitting position at 5-minute intervals.
32. Subject has a resting heart rate of <40 beats per minute or >100 beats per minute at screening.
33. Subject has an abnormal ECG at screening that is determined by the investigator to be clinically significant.
34. Male subject has a QTcF >450 ms or female subject has a QTcF >470 ms at screening or Day -1.
35. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hruby, PhD, Study Director — SIGA Chief Scientific Officer
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TPOXX
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TPOXX
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
Weight [Mean (Standard Deviation); unit: kg] | 138.13 (20.881)
Height [Mean (Standard Deviation); unit: cm] | 176.40 (9.649)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: Area under the plasma concentration vs. time curve (AUC) from time 0 to the last quantifiable measurement following Day 7 dose administration. Samples were collected before the AM dose (0 hour), at 0.5, 1, 2, 4, 6, 8, 12 (before the PM dose), 14, 16, 18, 20, and 24 hours (Day 8, 24 hours after the AM dose on Day 7), and on Day 9 (48 hours after the AM dose on Day 7).
Time Frame: Before the AM dose (0 hour), at 0.5, 1, 2, 4, 6, 8, 12 (before the PM dose), 14, 16, 18, 20, and 24 hours (Day 8, 24 hours after the AM dose on Day 7), and on Day 9 (48 hours after the AM dose on Day 7).
Population: PK population
Measure: Mean (Standard Error); unit: ng*h/mL
Arm/Group | TPOXX
Number analyzed (Participants) | 34
ng*h/mL | 29500 (26.0)

2. Primary Outcome: AUC0-24
Description: Area under the plasma concentration vs. time curve (AUC) from time 0 to the 24-hour time-point following Day 7 dose administration. Samples were collected before the AM dose (0 hour), at 0.5, 1, 2, 4, 6, 8, 12 (before the PM dose), 14, 16, 18, 20, and 24 hours (Day 8, 24 hours after the AM dose on Day 7).
Time Frame: Before the AM dose (0 hour), at 0.5, 1, 2, 4, 6, 8, 12 (before the PM dose), 14, 16, 18, 20, and 24 hours (Day 8, 24 hours after the AM dose on Day 7)
Population: PK population
Measure: Mean (Standard Error); unit: ng*h/mL
Arm/Group | TPOXX
Number analyzed (Participants) | 34
ng*h/mL | 20000 (23.0)

3. Primary Outcome: AUC0-inf
Description: AUC from time 0 extrapolated to infinity
Time Frame: Day 7
Population: PK population
Measure: Mean (Standard Error); unit: ng*h/mL
Arm/Group | TPOXX
Number analyzed (Participants) | 34
ng*h/mL | 33200 (27.8)

4. Primary Outcome: Cmax
Description: Maximum observed plasma drug concentration. Samples were collected before the AM dose (0 hour), at 0.5, 1, 2, 4, 6, 8, 12 (before the PM dose), 14, 16, 18, 20, and 24 hours (Day 8, 24 hours after the AM dose on Day 7), and on Day 9 (48 hours after the AM dose on Day 7). The median time to achieve Cmax was 4 hours post-dose.
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | TPOXX
Number analyzed (Participants) | 34
ng/mL | 1350 (29.0)

5. Primary Outcome: Tmax
Description: Time to reach Cmax
Time Frame: Day 7
Population: PK population
Measure: Median (Full Range); unit: h
Arm/Group | TPOXX
Number analyzed (Participants) | 34
h | 4.00 [2.00 to 11.95]

6. Primary Outcome: t1/2
Description: Terminal elimination half-life
Time Frame: Day 7
Population: PK population
Measure: Mean (Standard Error); unit: h
Arm/Group | TPOXX
Number analyzed (Participants) | 34
h | 12.9 (19.3)

7. Primary Outcome: CL/F
Description: Apparent total body clearance
Time Frame: Day 7
Population: PK population
Measure: Mean (Standard Error); unit: L/h
Arm/Group | TPOXX
Number analyzed (Participants) | 34
L/h | 64.8 (26.0)

8. Primary Outcome: Vd/F
Description: Apparent volume of distribution
Time Frame: Day 7
Population: PK population
Measure: Mean (Standard Error); unit: L
Arm/Group | TPOXX
Number analyzed (Participants) | 34
L | 1180 (29.9)

9. Primary Outcome: Ctrough
Description: Concentration observed prior to the next dose administration
Time Frame: Day 7
Population: PK population
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | TPOXX
Number analyzed (Participants) | 34
ng/mL | 617 (35.6)

10. Secondary Outcome: AEs as Assessed by CTCAE
Description: Number of subjects with AEs as assessed by CTCAE
Time Frame: 30 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | TPOXX
Number analyzed (Participants) | 34
participants | 12

11. Secondary Outcome: Subjects With at Least 1 AEs
Description: Number of subjects reported at least 1 adverse event
Time Frame: 30 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | TPOXX
Number analyzed (Participants) | 34
participants | 9

12. Secondary Outcome: Average Hemoglobin Concentration at Various Time Points; Mean (Standard Deviation)
Description: Table 14.3.2.1.1Summary of Actual Value and Change from Baseline in Hematology Safety Population Summary tables of observed values and changes from baseline: for hematology laboratory tests with numeric values for subjects in the Safety Population; to each scheduled post-baseline and changes in low, normal, high, and abnormal were summarized comparing the results at each scheduled post-baseline visit..
  Central laboratory reference ranges used for all clinical laboratory safety parameters
Time Frame: Baseline prior to dosing, 3 days post dose, 7 days post dose and 8 days post dose
Population: All subjects which were included in the safety population which is defined as all subjects who received at least one dose of TPOXX were included in this analysis.
Measure: Mean (Standard Deviation); unit: Hemoglobin (g/L)
Arm/Group | TPOXX
Number analyzed (Participants) | 34
Hemoglobin (g/L)
  Baseline | 138.0 (12.45)
  3 days post dose (Day 4) | 142.6 (14.43)
  7 days post dose (Day 8) | 142.0 (13.40)
  8 days post dose (Day 9) | 140.6 (13.35)

13. Secondary Outcome: Average Serum Chemistry at Various Time Points; Mean (Standard Deviation)
Description: Table 14.3.2.2.1 Laboratory Results - Serum Chemistry Safety Population Summary tables of observed values and changes from baseline: for serum chemistry laboratory tests with numeric values for subjects in the Safety Population; to each scheduled post-baseline and changes in low, normal, high, and abnormal were summarized comparing the results at each scheduled post-baseline.
  Central laboratory reference ranges used for all clinical laboratory safety parameters
Time Frame: Average Serum Chemistry at Baseline, 3 days post dose, 7 days post dose, and 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | TPOXX
Number analyzed (Participants) | 34
umol/L
  Bilirubin (umol/L) Baseline | 7.96 (3.339)
  Bilirubin (umol/L) 3 days post dose (Day 4) | 10.24 (3.760)
  Bilirubin (umol/L) 7 days post dose (Day 8) | 10.25 (3.393)
  Urate (umol/L) 3 days post dose (Day 4) | 406.0 (66.99)
  Urate (umol/L) 7 days post dose (Day 8) | 391.2 (65.17)
  Urate (umol/L) 8 days post dose (Day 9) | 391.5 (62.74)

14. Secondary Outcome: Average Urinalysis pH Values at Various Time Points:Day 9; Mean (Standard Deviation)
Description: Table 14.3.2.3.2 Laboratory Results - Urinalysis Safety Population Urinalysis laboratory tests with numeric values for subjects in the Safety Population; to each scheduled post-baseline and changes in low, normal, high, and abnormal were summarized comparing the results at each scheduled post-baseline visit.
  Central laboratory reference ranges used for all clinical laboratory safety parameters.
Time Frame: 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TPOXX
Number analyzed (Participants) | 34
pH | 5.93 (0.566)

15. Secondary Outcome: Average Systolic and Diastolic Blood Pressures at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.3.1.1 Vital Sign Results Safety Population
  Data listed shows the mean and standard deviation of systolic and diastolic blood pressure of 34 participants on day 9.
Time Frame: 9 days
Population: vital sign measurements values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TPOXX
Number analyzed (Participants) | 34
mmHg
  Systolic Blood Pressure (mmHg) 8 days post dose (Day 9) | 122.9 (11.41)
  Diastolic Blood Pressure (mmHg) 8 days post dose (Day 9) | 67.1 (8.91)

16. Secondary Outcome: Average Heart Rate at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.3.1.1 Vital Sign Results Safety Population
  Data listed shows the mean and standard deviation of heart rate of 34 participants on day 9.
Time Frame: 9 days
Population: Mean Heart Rate after dosing.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | TPOXX
Number analyzed (Participants) | 34
beats per minute | 77.0 (9.96)

17. Secondary Outcome: Average Respiratory Rate at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.3.1.1 Vital Sign Results Safety Population
  Data listed shows the mean and standard deviation of respiratory rates for 34 participants on day 9.
Time Frame: 9 days
Population: Mean Respiratory Rate after dosing.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | TPOXX
Number analyzed (Participants) | 34
breaths per minute | 14.8 (2.15)

18. Secondary Outcome: Average Body Temperature at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.3.1.1 Vital Sign Results Safety Population
  Data listed shows the mean and standard deviation of body temperatures for 34 participants on day 9.
Time Frame: 9 days
Population: Mean Body Temperature after dosing.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | TPOXX
Number analyzed (Participants) | 34
Celsius | 36.50 (0.281)

19. Secondary Outcome: Average 12-lead ECG at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.4.1.1 Electrocardiogram Results Safety Population Data listed shows the mean and standard deviation of 12 Lead EKG results for 34 participants on day 9.
Time Frame: 9 days
Population: Mean 12-lead ECG values after dosing.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TPOXX
Number analyzed (Participants) | 34
msec
  PR Interval, Aggregate (msec) 8 days post dose (Day 9) | 171.1 (20.43)
  QRS Duration, Aggregate (msec) 8 days post dose (Day 9) | 95.9 (10.38)

20. Secondary Outcome: Physical Examination at Baseline Compared to Physical Examination 9 Days Post Dose
Description: Listing 16.2.8.8 Physical Exam Safety Population
  Subjects were collated based on review of system and classified by assessment as "normal", "abnormal" or "assessments not done" on day 9.
Time Frame: 9 days
Population: Vital sign measurements, physical examination findings, and 12-lead ECG values after dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | TPOXX
Number analyzed (Participants) | 34
Participants
  8 days post dose (Day 9) Normal: Skin | 33
  8 days post dose (Day 9) Abnormal: Skin | 1
  8 days post dose (Day 9) Not Done: Skin | 0
  8 days post dose (Day 9) Normal: HEENT | 34
  8 days post dose (Day 9) Abnormal: HEENT | 0
  8 days post dose (Day 9) HEENT: Not Done | 0
  8 days post dose (Day 9) Normal: Pulmonary | 34
  8 days post dose (Day 9) Abnormal: Pulmonary | 0
  8 days post dose (Day 9) Not Done: Pulmonary | 0
  8 days post dose (Day 9) Normal: Cardiovascular | 34
  8 days post dose (Day 9) Abnormal: Cardiovascular | 0
  8 days post dose (Day 9) Not done: Cardiovascular | 0
  8 days post dose (Day 9) Abdomen: Normal | 34
  8 days post dose (Day 9) Abnormal: Abdomen | 0
  8 days post dose (Day 9) Not Done: Abdomen | 0
  8 days post dose (Day 9) Normal: Lymph Nodes | 34
  8 days post dose (Day 9) Abnormal: Lymph Nodes | 0
  8 days post dose (Day 9) Not Done: Lymph Nodes | 0
  8 days post dose (Day 9) Normal: Musculoskeletal | 33
  8 days post dose (Day 9) Abnormal: Musculoskeletal | 1
  8 days post dose (Day 9) Not Done: Musculoskeletal | 0
  8 days post dose (Day 9) Normal: Neurological System | 34
  8 days post dose (Day 9) Abnormal: Neurological System | 0
  8 days post dose (Day 9) Not Done: Neurological System | 0
  8 days post dose (Day 9) Normal: Other | 0
  8 days post dose (Day 9) Abnormal: Other | 0
  8 days post dose (Day 9) Not Done: Other | 34

21. Secondary Outcome: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase at Various Time Points Mean (Standard Deviation)
Description: as for outcome 13
Time Frame: Day 1 pre dose, 3 days, 7 days, and 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | TPOXX
Number analyzed (Participants) | 34
IU/L
  Alanine Aminotransferase (IU/L) Baseline | 21.8 (8.87)
  Alanine Aminotransferase (IU/L) 3 days post dose (Day 4) | 23.5 (11.84)
  Alanine Aminotransferase (IU/L) 7 days post dose (Day 8) | 25 (11.70)
  Alanine Aminotransferase (I/UL) 8 days post dose (Day 9) | 25.6 (12.21)
  Alk Phosphate (IU/L) Baseline | 64.9 (20.51)
  Alk Phosphate (IU/L)3 days post dose (Day 4) | 61.0 (19.42)
  Alk Phosphate (IU/L) 7 days post dose (Day 8) | 66.9 (20.90)
  Alk Phosphate (IU/L) 8 days post dose (Day 9) | 67.4 (20.56)
  Aspartate Aminotransferase (IU/L) Baseline | 17.6 (4.63)
  Aspartate Aminotransferase (IU/L) 3 days post dose (Day 4) | 18.2 (5.69)
  Aspartate Aminotransferase (IU/L) 7 days post dose (Day 8) | 17.9 (4.49)
  Aspartate Aminotransferase (IU/L) 8 days post dose (Day 9) | 18.3 (4.46)
  Gamma Glutamyl Transferase (IU/L) Baseline | 27.4 (12.89)
  Gamma Glutamyl Transferase (IU/L) 3 days post dose (Day 4) | 27.6 (12.81)
  Gamma Glutamyl Transferase (IU/L) 7 days post dose (Day 8) | 28.6 (12.91)
  Gamma Glutamyl Transferase (IU/L) 8 days post dose (Day 9) | 28.6 (13.01)
  Lactate Dehydrogenase (IU/L) Baseline | 159.2 (33.00)
  Lactate Dehydrogenase (IU/L) 3 days post dose (Day 4) | 147.8 (34.86)
  Lactate Dehydrogenase (IU/L) 7 days post dose (Day 8) | 142.9 (33.20)
  Lactate Dehydrogenase (IU/L) 8 days post dose (Day 9) | 148.1 (33.20)

22. Secondary Outcome: Albumin, Globulin, and Protein at Various Time Points Mean (Standard Deviation)
Description: as for outcome 13
Time Frame: Day 1 pre dose, 3 days post dose, 7 days post dose and 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | TPOXX
Number analyzed (Participants) | 34
g/L
  Albumin (g/L) Baseline | 42.4 (2.78)
  Albumin (g/L) 3 days post dose (Day 4) | 43.4 (3.35)
  Albumin (g/L) 7 days post dose (Day 8) | 43.5 (2.61)
  Albumin (g/L)8 days post dose (Day 9) | 44.2 (2.73)
  Globulin (g/L) Baseline | 27.3 (3.87)
  Globulin (g/L) 3 days post dose (Day 4) | 29.1 (3.53)
  Globulin (g/L) 7 days post dose (Day 8) | 28.6 (3.78)
  Globulin (g/L) 8 days post dose (Day 9) | 28.9 (3.81)
  Protein (g/L) Baseline | 69.7 (5.13)
  Protein (g/L) 3 days post dose (Day 4) | 72.4 (5.16)
  Protein (g/L) 7 days post dose (Day 8) | 72.1 (4.46)
  Protein (g/L) 8 days post dose (Day 9) | 73.1 (4.90)

23. Secondary Outcome: Average Serum Chemistry at Various Time Points; Mean (Standard Deviation)
Description: as for outcome 13
Time Frame: Day 1 pre dose, 3, 7, and 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | TPOXX
Number analyzed (Participants) | 34
mmol/L
  Anion Gap (mmol/L) Baseline | 10.6 (1.5)
  Anion Gap (mmol/L) 3 days post dose (Day 4) | 10.4 (2.15)
  Anion Gap (mmol/L) 7 days post dose (Day 8) | 10.6 (1.65)
  Anion Gap (mmol/L) 8 days post dose (Day 9) | 10.3 (1.38)
  Blood Urea Nitrogen (mmol/L) Baseline | 4.415 (1.05)
  Blood Urea Nitrogen (mmol/L) 3 days post dose (Day 4) | 4.231 (0.7147)
  Blood Urea Nitrogen (mmol/L) 7 days post dose (Day 8) | 4.091 (0.6397)
  Blood Urea Nitrogen (mmol/L) 8 days post dose (Day 9) | 4.346 (0.6745)
  Calcium (mmol/L) Baseline | 2.304 (0.0980)
  Calcium (mmol/L) 3 days post dose (Day 4) | 2.360 (0.0921)
  Calcium (mmol/L) 7 days post dose (Day 8) | 2.397 (0.0921)
  Calcium (mmol/L) 8 days post dose (Day 9) | 2.348 (0.0852)
  Carbon Dioxide (mmol/L) Baseline | 29.2 (1.47)
  Carbon Dioxide (mmol/L) 3 days post dose (Day 4) | 29.5 (2.02)
  Carbon Dioxide (mmol/L) 7 days post dose (Day 8) | 29.8 (1.55)
  Carbon Dioxide (mmol/L) 8 days post dose (Day 9) | 29.4 (1.78)
  Chloride (mmol/L) Baseline | 102.6 (1.48)
  Chloride (mmol/L) 3 days post dose (Day 4) | 103.0 (1.55)
  Chloride (mmol/L) 7 days post dose (Day 8) | 102.2 (1.68)
  Chloride (mmol/L) 8 days post dose (Day 9) | 101.9 (1.56)
  Glucose (mmol/L) Baseline | 5.401 (0.4533)
  Glucose (mmol/L) 3 days post dose (Day 4) | 5.276 (0.4118)
  Glucose (mmol/L) 7 days post dose (Day 8) | 5.088 (0.4252)
  Glucose (mmol/L) 8 days post dose (Day 9) | 5.169 (0.3683)
  Phosphate (mmol/L) Baseline | 1.115 (0.1642)
  Phosphate (mmol/L) 3 days post dose (Day 4) | 1.246 (0.1668)
  Phosphate (mmol/L) 7 days post dose (Day 8) | 1.282 (0.1600)
  Phosphate (mmol/L) 8 days post dose (Day 9) | 1.104 (0.1363)
  Potassium (mmol/L) Baseline | 4.12 (0.263)
  Potassium (mmol/L) 3 days post dose (Day 4) | 4.15 (0.230)
  Potassium (mmol/L) 7 days post dose (Day 8) | 4.17 (0.244)
  Potassium (mmol/L) 8 days post dose (Day 9) | 4.13 (0.303)
  Sodium (mmol/L) Baseline | 138.2 (1.57)
  Sodium (mmol/L) 3 days post dose (Day 4) | 138.9 (1.62)
  Sodium (mmol/L) 7 days post dose (Day 8) | 138.5 (1.69)
  Sodium (mmol/L) 8 days post dose (Day 9) | 137.4 (1.88)

24. Secondary Outcome: Urobilinogen (Umol/dl) 8 Days Post Dose (Day 9); Mean (Standard Deviation)
Description: Table 14.3.2.3.2 Laboratory Results - Urinalysis Safety Population Summary tables of observed values and changes from baseline: for urinalysis laboratory tests with numeric values for subjects in the Safety Population; to each scheduled post-baseline and changes in low, normal, high, and abnormal were summarized comparing the results at each scheduled post-baseline visit.
  Central laboratory reference ranges used for all clinical laboratory safety parameters.
Time Frame: 8 days post dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: umol/dl
Arm/Group | TPOXX
Number analyzed (Participants) | 34
umol/dl | 1.0196 (0.00640)

25. Secondary Outcome: 12-lead ECG Heart Rate at 9 Day Time Point; Mean (Standard Deviation)
Description: Table 14.3.4.1.1 Electrocardiogram Results Safety Population Data listed shows the mean and standard deviation of 12 Lead EKG heart rate for 34 participants on day 9.
Time Frame: 9 days
Population: Mean 12-lead ECG values after dosing.
Measure: Mean (Standard Deviation); unit: bats per minute
Arm/Group | TPOXX
Number analyzed (Participants) | 34
bats per minute | 71.0 (9.66)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study drug until study Day 37 (+2 days).
Description: An AE is any event or any untoward medical occurrence, including those AEs that result from dosing error, which may present during administration of a study drug, or during a reasonable follow-up period, and which does not necessarily have a causal relationship with this treatment.
Arm/Group | TPOXX
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 12/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPOXX (N=34)
Headache (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Scleral hyperaemia (Eye disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Palate injury (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT04392739/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT04392739/SAP_001.pdf